CLINICAL TRIAL: NCT02376894
Title: An Epidemiological Survey of Cancer-related Fatigue Among Taiwanese Cancer Patients
Status: Completed | Type: Observational
Sponsor: Taiwan Cancer Palliative Medicine (Other)
Collaborators: National Taiwan University Hospital (Other); Shin Kong Wu Ho-Su Memorial Hospital (Other); Tri-Service General Hospital (Other); Changhua Christian Hospital (Other); National Cheng-Kung University Hospital (Other); Chung Shan Medical University (Other); Kaohsiung Veterans General Hospital. (Other); Taipei Veterans General Hospital, Taiwan (Other Government); Taipei Medical University Hospital (Other); Taipei Medical University Shuang Ho Hospital (Other); Taipei Medical University WanFang Hospital (Other); China Medical University Hospital (Other); Mackay Memorial Hospital (Other); Far Eastern Memorial Hospital (Other); Chang Gung Memorial Hospital (Other); Chiayi Christian Hospital (Other); Taipei Tzu Chi Hospital, Buddhist Tzu Chi Medical Foundation (Other); Taichung Tzu Chi Hospital (Other); Chi Mei Medical Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: CRF-TSCPM01
Record Dates: First submitted 2015-02-25; First posted 2015-03-03 (Estimated); Last update posted 2018-01-10 (Actual); Status verified 2018-01

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
The aim of this study is to examine the prevalence, severity, impacts and managements of CRF among Taiwanese cancer patients.

DETAILED DESCRIPTION:
The cross-sectional survey is conducted at oncology inpatients unit and outpatients clinics of hospitals in Taiwan. Furthermore, the results will elucidate not only the epidemiology of CRF in Taiwan, but will supply physicians with more understanding about CRF, and help them to enhance the quality on cancer care to being perfected in the future.

ELIGIBILITY:
Inclusion Criteria:

* (1) Patients who signed the informed consent form
* (2) The age of eligible patients should be > 20 years old.
* (3) Inpatients or outpatients who have been given a diagnosis of cancer
* (4) Able to communicate verbally and completely fill out the questionnaires

Exclusion Criteria:

* Patients who have been given a diagnosis of cognitive impairment are unable to complete the questionnaires

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: cancer patient
Sampling Method: Non-Probability Sample
Enrollment: 1211 (Actual)
Dates: Start 2015-02 (Actual); Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Cancer-related fatigue evaluation | 30 minuts
  ICD-10 Fatigue Criteria,Brief Fatigue Inventory-Taiwan Form
Symptoms and Quality of Life Assessments | 15 minutes
  FACT-G7

CONTACTS AND LOCATIONS:
Locations (1):
- Taipei Medical University Hospital, Taipei, Taiwan